CLINICAL TRIAL: NCT03361969
Title: A Double-blind, Randomised, Placebo-controlled, Multi-center Study to Evaluate Effects of Estetrol on Testosterone Suppression and Quality of Life in Prostate Cancer Patients Treated With an LHRH Agonist.
Brief Title: Evaluation of Effects of Estetrol on Testosterone Suppression and Quality of Life in Prostate Cancer Patients Treated With an LHRH Agonist.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pantarhei Oncology B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR3109
Record Dates: First submitted 2017-11-21; First posted 2017-12-05 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Prostatic Neoplasm
Keywords: quality of life; hot flushes; prostate cancer; testosterone
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes | interventions — Estetrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- estetrol (Active Comparator)
  Interventions: Drug: Estetrol
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Estetrol — estetrol formulated in tablets
  Arms: estetrol
Drug: Placebo Oral Tablet — placebo tablets
  Arms: placebo

SUMMARY:
This is a phase IIa, double-blind, randomised, placebo-controlled, multi-center study to evaluate the effects of estetrol on testosterone suppression and quality of life in prostate cancer patients treated with an LHRH agonist. Patients will be treated with estetrol or placebo for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with prostate cancer, qualifying for treatment with a LHRH agonist;
* Age ≥ 18 years;
* Body mass index (BMI) between ≥ 18.0 and ≤ 35.0 kg/m2 (inclusive);
* Reasonable physical and mental health as judged by the Investigator determined by physical examination, clinical laboratory assessments and vital signs;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1;
* Life expectancy of at least 2 years.

Exclusion Criteria:

* Current or prior (during the last 12 months) hormonal therapy, immunotherapy or chemotherapy for prostate cancer. Allowed are 14 days concomitant treatment with an anti-androgen to prevent the flare-up, radiotherapy and low dose radiation to prevent gynecomastia;
* History of deep vein thrombosis, pulmonary embolism, or cerebrovascular accident. However, patients with such history using anticoagulants for ≥ 6 months are eligible for the study provided anticoagulant treatment is continued throughout the whole study;
* History of myocardial infarction or a coronary vascular procedure (e.g. percutaneous coronary intervention, coronary artery bypass graft). However, patients with such history using anticoagulants for ≥ 6 months are eligible for the study provided anticoagulant treatment is continued throughout the whole study;
* Patients who have unstable angina or clinical congestive heart failure;
* A defect in the blood coagulation system, assessed at screening: deficiencies in AT-III, protein C and protein S and elevated factor VIII;
* Mutation in coagulation factor II and/or positive for factor V Leiden, assessed at screening;
* Diabetes mellitus with poor glycaemic control in the past 6 months (haemoglobin A1c (HbA1c) above 7.5%);
* Known primary hyperlipidaemias (Fredrickson);
* Disturbance of liver function: cholestatic jaundice, a history of jaundice due to previous estrogen use, Rotor syndrome and Dubin-Johnson syndrome;
* Known porphyria;
* Uncontrolled hypertension, i.e. systolic blood pressure 160 mmHg and/or diastolic blood pressure 100 mmHg in the last 6 months with or without medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Difference in total testosterone levels between treatment groups | 168 days
  Serum concentrations of total testosterone will be listed and summarized descriptively by treatment group. Nadir and time to nadir will be described using summary statistics.
Difference in free testosterone levels between treatment groups | 168 days
  Serum concentrations of free testosterone will be listed and summarized descriptively by treatment group. Nadir and time to nadir will be described using summary statistics.
Difference in mean daily hot flushes score between treatment groups | 168 days
  The number and severity in hot flushes will be assessed by means of a diary in which the patients records his hot flushes for 7 days.

SECONDARY OUTCOMES:
Change from baseline in endocrine parameters, adrenal androgen, dihydrotestosterone (DHT) and Sex Hormone Binding Globulin (SHBG) | 168 days
  Effects on endocrine parameters (Luteinising Hormone (LH), Follicle Stimulating Hormone (FSH) and Estradiol (E2), adrenal androgens (Dehydroepiandrosterone sulfate (DHEAS)), dihydrotestosterone (DHT) and SHBG will be evaluated. Actual values at baseline and at the scheduled visits, as well as change from baseline values at the post-baseline visits will be described using summary statistics and graphs. Difference between the treatment groups will be evaluated.
Change from baseline in prostate-specific antigen (PSA) response | 168 days
  Effects on PSA response will be evaluated. Actual values at baseline and at the scheduled visits, as well as change from baseline and percentage change from baseline values at the post-baseline visits will be described using summary statistics and graphs. Nadir and time to nadir will be described using summary statistics. Difference between the treatment groups will be evaluated.
Questionnaire on Quality of Life | 168 days
  Effects on FACT-P questionnaire will be evaluated. FACT-P includes a 27-item "core" quality of life measure (FACT-G) grouped into 4 sub-scales: physical, social/family, emotional, and functional well-being. The prostate cancer-specific subscale contains an additional 12 items; 10 of which are prostate cancer specific physical problems. Items are rated on a 5-item Likert scale, from 0, "not at all", to 4, "very much". Total range of scores is from 0 - 156. Higher scores indicate higher degree of functioning and better quality of life.
  Total FACT-P scores, FACT-P general health subscale score (FACT-G) total score and all FACT-P subscale scores will be described at the scheduled visits using summary statistics and graphs. Differences between the treatment groups will be evaluated.
Change from baseline in lipids | 168 days
  Effects on total cholesterol, triglycerides, High Density Lipoprotein (HDL) cholesterol and Low Density Lipoprotein (LDL) cholesterol will be evaluated. Actual values at baseline and at the schedule visits as well as change from baseline values at the post-baseline visits will be described using summary statistics and graphs. Differences between the treatment groups will be evaluated.
Change from baseline in bone turnover markers | 168 days
  Effects on bone turnover markers osteocalcin and type I collagen telopeptide (CTX-1) will be evaluated. Actual values at baseline and at the schedule visits as well as change from baseline values at the post-baseline visits will be described using summary statistics and graphs. Differences between the treatment groups will be evaluated.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Andros Men's Health Institutes, Arnhem, Gelderland
  - Noord West Ziekenhuis, Alkmaar
  - St Antonius Ziekenhuis, Nieuwegein
  - CWZ, Nijmegen
  - Antonius Ziekenhuis, Sneek
  - Isala Zwolle, Zwolle